CLINICAL TRIAL: NCT00804011
Title: Automatic Tube Compensation Versus Pressure Support in Weaning Patients With Severe Neurotoxic Snake Envenoming
Brief Title: Automatic Tube Compensation (ATC) for Weaning Patients With Severe Neurotoxic Snake Envenoming
Acronym: ATC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Dept of Pulmonary Medicine, PGIMER, Chandigarh (Unknown)
Responsible Party: Dr Ritesh Agarwal, PGIMER, India
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS/486/Res/507
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Snake Bite; Weaning; Mechanical Ventilation
Keywords: Snakebite; Weaning; Mechanical ventilation
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Automatic tube compensation plus pressure support
  Interventions: Other: ATC
- 2 (Active Comparator): Pressure support alone
  Interventions: Other: PSV

INTERVENTIONS:
Other: ATC — Automatic tube compensation
  Other Names: Automatic tube compensation
  Arms: 1
Other: PSV — Pressure support ventilation
  Other Names: Pressure support ventilation
  Arms: 2

SUMMARY:
In the mechanically ventilated patient, the single greatest cause of imposed work of breathing is the resistance caused by the endotracheal tube. Commonly used maneuvers to overcome this resistance include the use of continuous positive airway pressure or pressure support.However, a new mode of ventilatory support called automatic tube compensation (ATC) delivers exactly the amount of pressure necessary to overcome the resistive load imposed by the endotracheal tube for the flow measured at the time (so called variable pressure support).

The aim of this study is to evaluate whether a combination of pressure support with automatic tube compensation is superior to PS alone in weaning patients with severe neurotoxic snake envenoming.

DETAILED DESCRIPTION:
Snake envenoming is a common medical emergency encountered in the tropical countries, and an estimated 35,000 to 50,000 people die of snake bite every year in India. The bites of Elapid snakes cause predominantly neurotoxicity, which manifests as paralysis of the muscles of the eyes, tongue, throat and respiration, leading to respiratory failure, and if untreated death. The management of these patients includes ventilatory support and administration of snake anti-venom (SAV). Respiratory failure, requiring mechanical ventilatory support, is a frequent cause for admission to the intensive care unit (ICU).

Mechanical ventilation is a life-saving intervention and once there is improvement of the underlying indication for mechanical ventilation, it can be withdrawn abruptly in the majority. However, approximately 20-30% of patients still require gradual discontinuation i.e. weaning. This process is not only difficult in patients with chronic respiratory diseases and neuromuscular disorders like neurotoxic snake bite, but is also associated with significant complications like pneumonia, prolonged ICU stay and even mortality, especially in those with persistent weaning failure.

In the mechanically ventilated patient, it has long been recognized that the single greatest cause of imposed work of breathing (WOB) is the resistance caused by the endotracheal tube (ETT). Commonly used maneuvers to overcome the ETT resistance include the use of continuous positive airway pressure (CPAP) or pressure support (PS). However, a new mode of ventilatory support called automatic tube compensation (ATC) delivers exactly the amount of pressure necessary to overcome the resistive load imposed by the endotracheal tube for the flow measured at the time (so called variable pressure support). This mode theoretically can decrease weaning duration and increase the probability of successful extubation by decreasing the WOB.

Recently, we have reported our ICU data of 55 patients of severe neurotoxic snake envenoming in which we evaluated if usage of a higher dosage of SAV offered any significant clinical advantage over a lower dose, and found no difference between the high-dose and low-dose groups. The aim of this study is to evaluate whether a combination of PS with ATC is superior to PS alone in weaning patients with severe neurotoxic snake envenoming.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe neurotoxic snake envenoming (defined as requirement of mechanical ventilation for ventilatory failure) will be included in the study. - Snake envenoming will be diagnosed on the history of snakebite, presence of fang marks, presence of local manifestations such as swelling, cellulitis, blister formation; or if the dead snake is brought for identification.
* Significant improvement in the neuroparalysis with improvement in grade of power to at least MRC 3
* Normal sensorium
* Minimal suction requirements (less than thrice in the eight hours preceding the assessment
* No requirement for any vasoactive drugs
* No sedation (vi) core temperature less than 38.0°C
* Hemoglobin more than 9 gm/dL (viii) systolic blood pressure more than 90 mm Hg
* Overall physician assessment whether the patient is fit for weaning.

Exclusion Criteria:

* If they do not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-07; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Duration of weaning | 6 month

SECONDARY OUTCOMES:
ICU stay | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, MD, DM, FCCP, Principal Investigator — PGIMER, INDIA; Ashutosh N Aggarwal, MD, DM, FCCP, Study Chair — PGIMER, INDIA
Locations (1):
- Department of Pulmonary Medicine, Chandigarh, Uttarakhand, India